CLINICAL TRIAL: NCT03608254
Title: Acute Effects of Watermelon on Vascular Function and Serum Lycopene
Status: Completed | Type: Observational
Sponsor: University of Alabama, Tuscaloosa (Other)
Responsible Party: Principal Investigator, Amy Ellis, Assistant Professor, University of Alabama, Tuscaloosa
Other Study IDs: 15-07-95
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Results first posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2021-12

CONDITIONS: Vascular Health of Postmenopausal Women

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Banked serum will be stored at -80 degrees C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 100% watermelon juice — Participants consumed a one-time dose of 100% watermelon juice. Blood was sampled before and 2 hours after ingestion. Blood pressure and brachial artery flow-mediated dilation were measured before and 2 hours after ingestion.

SUMMARY:
This study aimed to examine the effects of a one-time dose of 100% watermelon juice on circulating lycopene levels and measures of vascular health among a cohort of postmenopausal women.

DETAILED DESCRIPTION:
Purpose and Objectives Arterial stiffness and endothelial dysfunction are early independent predictors of cardiovascular disease (CVD), the leading cause of death for women ages 60 and older in the United States. It is well-known that age-related decreases in vascular function are partially due to increases in oxidative stress and inflammation. In attempts to combat CVD, previous studies have investigated provision of isolated food compounds in supplement form. For example, purified lycopene has been shown to decrease oxidative stress, and our previous work supports the supplemental use of glutamine and arginine powders for improving vascular endothelial function of older adults. Watermelon is among the greatest plant sources of arginine and glutamine, and it is one of the richest sources of lycopene. However, clinical studies evaluating the whole food have not been done.

According to the Healthy Eating Index, only 27% of women ages 60 and older meet the daily dietary recommendations for 2.5 fruit servings. Likewise, although no Recommended Dietary Allowance for lycopene exists, this age group consumes less lycopene daily than is provided in one serving of watermelon. While reasons for poor fruit intake among older adults are multifactorial, difficulty chewing and inability to prepare fresh foods in the home environment have been noted as significant barriers to fresh fruit and vegetable intake. Of note, a previous systematic review suggests that 100% fruit and vegetable juices may be practical vehicles for improving intake of antioxidant nutrients among older adults. The provision of 100% watermelon juice to older adult women represents a practical, innovative approach to increase consumption of a food containing multiple components that may act in synergy to improve vascular function. Therefore, the purpose of this study is to investigate the effects of a one-time serving of 100% watermelon juice on blood vessel function and serum lycopene.

Specific Aims

The specific aims of this study are to:

1. To determine whether consumption of a 12-ounce serving of 100% watermelon juice by non-obese women ages 60-75 will result in increased levels of serum lycopene.

   Hypotheses: Acute supplementation with 100% watermelon juice will result in increased serum lycopene.
2. To determine whether consumption of a 12-ounce serving of 100% watermelon juice by non-obese women ages 60-75 will result in improved vascular endothelial function as assessed by flow-mediated dilation (FMD) and decreased arterial stiffness as assessed by pulse wave analysis (PWA).

Hypotheses: Acute supplementation with 100% watermelon juice will result in improved vascular endothelial function and decreased arterial stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.5 - 29.9 kg/m2 (non-obese)
* Ambulatory
* Postmenopausal female
* Ages 65-70 years

Exclusion Criteria:

* Food allergy to watermelon
* Diagnosis of phenylketonuria
* History of hypotension, chronic uncontrolled hypertension, chronic kidney disease, diabetes, previous cardiac events or procedures,
* Smoking or other tobacco use
* Use of anticoagulant medications, cholesterol-lowering medications, vasodilatory dietary supplements (garlic, fish oil), or dietary supplements containing lycopene, ascorbic acid, L-glutamine, L-arginine, or L-citrulline
* Weight change > 10% in the previous six months

Ages: 65 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling postmenopausal women
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2016-12-08 (Actual); Study Completion 2016-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Ellis, PhD, RD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Tuscaloosa, Alabama, United States

REFERENCES:
- [Derived] Ellis AC, Dudenbostel T, Crowe-White K. Watermelon Juice: a Novel Functional Food to Increase Circulating Lycopene in Older Adult Women. Plant Foods Hum Nutr. 2019 Jun;74(2):200-203. doi: 10.1007/s11130-019-00719-9. PMID 30756297

RESULTS

PARTICIPANT FLOW:
Groups:
- Watermelon Juice: All participants consumed 12 ounces of 100% watermelon juice. Blood samples were taken, and flow-mediated dilation was measured before consumption of the juice and two hours afterward.
Period: Overall Study
Arm/Group | Watermelon Juice
Started | 11
Completed | 8
Not Completed | 3
Not completed — Blood sampling was not completed for 2 participants. | 2
Not completed — One participant chose not to consume the entire 12-ounce dose of watermelon juice. | 1

BASELINE CHARACTERISTICS:
Population: Eleven participants were consented to participate in the cross-sectional study. Eight participants completed all study measures. Blood sampling was not possible for two participants, and one participant did not consume the total test dose of watermelon juice.
Arm/Group | Watermelon Juice
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.73 (2.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Serum lycopene [Mean (Standard Deviation); unit: umol/L] | 1.48 (1.07)
Flow-mediated dilation (FMD) [Mean (Standard Deviation); unit: percent change in diameter] — FMD uses ultrasound technology to quantify changes in brachial artery diameter in response to hyperemia. A blood pressure cuff was placed distal to the brachial artery of the right arm with the participant supine and rested. Pre-inflation diameter was recorded for one minute, and the cuff was inflated to 50 mmHg above resting SBP for five minutes. Then, images were recorded for 120 seconds after cuff deflation. Peak diameter was determined as an average of the five highest measurements over five seconds post-deflation. FMD was expressed as the percentage increase in peak diameter.
  percent change in diameter | 9.93 (6.09)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Circulating Lycopene Levels
Description: On the testing day, participants reported to the clinic following a 10-hour overnight fast. Blood samples were obtained by standard venipuncture at baseline and two hours after ingestion of a 360 ml dose of 100% pasteurized watermelon juice in order to determine change in serum lycopene levels.
Time Frame: 2 hours post-ingestion
Population: Eleven participants provided consent for the cross-sectional study. Blood sampling was not possible for two participants, and one participant did not consume the entire 12-ounce dose of juice.
Measure: Mean (Standard Deviation); unit: umol/L
Groups:
- Watermelon Juice: Participants consumed 12 ounces of 100% watermelon juice. Blood samples were taken, and flow-mediated dilation was measured before consumption of the juice and two hours afterward.
Arm/Group | Watermelon Juice
Number analyzed (Participants) | 8
umol/L | 2.85 (0.66)

2. Secondary Outcome: Change From Baseline in Endothelial-dependent Vasodilation
Description: Brachial artery flow-mediated dilation (FMD) was used to assess endothelial-dependent vasodilation. FMD uses ultrasound technology to quantify changes in brachial artery diameter in response to hyperemia. A blood pressure cuff was placed distal to the brachial artery of the right arm with the participant supine and rested. Pre-inflation diameter was recorded for one minute, and the cuff was inflated to 50 mmHg above resting SBP for five minutes. Then, images were recorded for 120 seconds after cuff deflation. Peak diameter was determined as an average of the five highest measurements over five seconds post-deflation. FMD was expressed as the percentage increase in peak diameter. FMD measurements were taken at baseline and 2 hours after ingestion of the 100% watermelon juice. The outcome measure reflects change in FMD from baseline to 2 hours post-ingestion.
Time Frame: 2 hours post-ingestion
Population: One participant did not consume the entire 12-ounce dose of juice.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Watermelon Juice
Number analyzed (Participants) | 10
percent change from baseline | 2.33 (7.33)

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events the day they participated in the study.
Arm/Group | Watermelon Juice
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No